CLINICAL TRIAL: NCT02628795
Title: Overcoming TWEAK Signaling to Restore Muscle and Mobility After Joint Replacement
Acronym: TWEAK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Marcas M. Bamman, PhD, Professor and Director, UAB Center for Exercise Medicine, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01HD084124 (NIH); R01HD084124 (NIH)
Record Dates: First submitted 2015-08-05; First posted 2015-12-11 (Estimated); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Osteoarthritis
Keywords: total hip arthroplasty; total knee arthroplasty
MeSH Terms: conditions — Osteoarthritis | interventions — Hypoxanthine Phosphoribosyltransferase

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PRT + FM (Experimental): Progressive resistance training + functional mobility training 3 d/wk x 16 wk
  Interventions: Behavioral: PRT + FM; Other: Usual Care
- Usual Care (Active Comparator): Post-surgical usual care including physical therapy
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: PRT + FM — Supervised progressive resistance training + functional mobility training (PRT+FM) 3 days per week for 16 weeks post-surgery.
  Arms: PRT + FM
Other: Usual Care — Post-surgical usual care activities including any prescribed physical therapy

SUMMARY:
This single-blind, randomized, controlled trial is designed to test the effect of an intensive, 16 week exercise rehabilitation program (progressive resistance training + functional mobility training) vs. usual care on restoration of muscle mass and mobility after total hip (THA) or knee (TKA) arthroplasty in men and women with end-stage osteoarthritis. The molecular basis underlying the trial is the presence of significant muscle inflammation susceptibility in many of these individuals, and the expectation that the more intensive intervention will overcome this inflammatory burden to facilitate recovery.

DETAILED DESCRIPTION:
While elective total hip (THA) and knee (TKA) arthroplasty relieve pain and improve mobility function for thousands with end-stage osteoarthritis (OA), up to 35% endure persistent muscle atrophy and mobility limitations for several years that impact life quality, increase morbidity, and burden the healthcare system. Given that THA/TKA volumes are increasing exponentially with >1.1 million in the US annually, refractory mobility impairment is a major public health problem. Together, the available data raise two important knowledge gaps in THA/TKA rehabilitation: (i) poorly understood factors that limit responsiveness of a large number of patients to current usual care; and (ii) the absence of rehabilitation programs proven to overcome these limitations. The proposed project is designed to fill these gaps. The investigators' fundamental tenet is that restoration of mobility function following THA/TKA requires: (i) regeneration of surgically damaged muscle; and (ii) regrowth of muscles that have atrophied over years of OA and limited usage. The investigators suggest a major cause of muscle regeneration impairment in some individuals is what the investigators identified as muscle inflammation susceptibility (MuIS) - hyperactive inflammatory signaling in muscle of MuIS(+) individuals despite no systemic inflammation - which also manifests in isolated primary satellite cells and inhibits myogenesis in vitro, indicative of a true cellular phenotype beyond the niche. The investigators' preliminary findings in THA/TKA patients strongly suggest the tumor necrosis factor-like weak inducer of apoptosis (TWEAK) signaling pathway may be central to MuIS and impaired THA/TKA recovery, as high perioperative muscle TWEAK signaling in the ipsilateral thigh was the most sensitive indicator of impaired muscle protein synthesis and failed strength recovery after 8 wk of usual care. Progressive resistance exercise training (PRT) is a putative anabolic intervention that the investigators find consistently increases muscle mass to meet healthy standards in atrophied and mobility-impaired adults, by activating muscle protein synthesis and the myogenic activity of muscle satellite cells. Together, these findings raise the central hypothesis that PRT plus adjunctive functional mobility training (PRT+FM) after THA/TKA will more effectively restore muscle mass and mobility function to healthy standards than usual care and, because MuIS(+) are predicted to suffer failed muscle recovery and persistent dismobility under usual care, the impact of PRT+FM will be greatest in MuIS(+). The investigators will thoroughly test this hypothesis in a randomized controlled trial of 88 THA/TKA patients with the following aims. Aim 1: To determine the effects of 16 wk of PRT+FM vs. usual care after elective THA/TKA on muscle mass, performance, and mobility function. Aim 2: To determine whether MuIS status modifies the effects of PRT+FM or usual care after THA/TKA. Cellular and molecular mechanisms of muscle mass regulation will be studied in detail. Aim 3. To determine the long-term impact of 16 wk PRT+FM by re-assessing outcomes at 6 mo and 1 y. The investigators fully expect the novel findings to lead a paradigm shift in THA/TKA rehabilitation that will have a profound impact on a growing segment of the population.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages 40 and 80 y.

  * Scheduled to undergo elective total hip or knee replacement specifically for the surgical indication of end-stage osteoarthritis.
  * First-time hip or knee replacement.
  * Capable of providing informed consent (cognitively intact if consenting to surgery).

Exclusion Criteria:

* Any surgical indication other than first-time total joint replacement specifically for end-stage osteoarthritis.

  * Bilateral knee/ hip replacement
  * History of alcoholism or liver disease.
  * Any history of hypo- or hyper-coagulation disorders including subjects taking Coumadin.
  * Any individual with end-stage disease and/or a life expectancy less than one year.
  * Pregnancy.
  * Lactating Women.
  * Neurological, musculoskeletal, or other disorder that would preclude them from completing the exercise training intervention and all performance tests.
  * Uncontrolled hypertension, unstable or exercise-induced angina pectoris or myocardial ischemia, congestive heart failure.
  * Uncontrolled diabetes mellitus.
  * Any other condition or events considered exclusionary by the PIs and/or physician Co-Is.
  * Lidocaine allergy (1% lidocaine is the local anesthetic used during the muscle biopsy procedure).
  * Phenylketonuria (phenylalanine tracer for metabolic studies).
  * Currently receiving androgen (e.g., testosterone) or anabolic (e.g., growth hormone (GH), insulin-like growth factor-I (IGF-I)) therapy.
  * Body mass index ≥ 35.
  * History of lower body progressive resistance training within the past year.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Change in unilateral (surgical) thigh muscle mass (unit of measure = grams) | Pre-surgery to 16 weeks post-surgery
  Primary muscle mass outcome of Aim 1
Change in unilateral (surgical) knee extension power (unit of measure = watts) | Pre-surgery to 16 weeks post-surgery
  Primary functional outcome of Aim 1
Change in short physical performance battery (SPPB) (unit of measure = score) | From 16 weeks post-surgery to 26 and 52 weeks post-surgery
  Primary outcome of Aim 3
Muscle inflammation susceptibility (MuIS) status (unit of measure = relative value) | At the time of surgery
  Primary outcome of Aim 2: Muscle inflammation susceptibility (MuIS) defined by TWEAK receptor gene expression

SECONDARY OUTCOMES:
Change in muscle fiber size (unit of measure = micrometers squared) | From the time of surgery to 16 weeks post-surgery
Change in unilateral (surgical) knee extension isometric strength (unit of measure = Newton-meters) | Pre-surgery to 16 weeks post-surgery
Change in maximum 10-meter gait speed (unit of measure = meters per second) | Pre-surgery to 16 weeks post-surgery

OTHER OUTCOMES:
Change in free-living physical activity (unit of measure = steps per day) | Pre-surgery to 8, 16, 26, and 52 weeks post-surgery
  Via wearable technology (i.e. step counter)
Change in self-reported health status (unit of measure = score) | Pre-surgery to 1, 8, 16, 26, and 52 weeks post-surgery
  Via Short Form-36v2 Health Survey (SF-36v2)
Change in cellular and molecular markers (unit of measure = arbitrary units) | From the time of surgery to 16 weeks post-surgery
  Experiments using muscle tissue and primary muscle satellite cells collected from surgical and contralateral limbs.
Change in fatigue (unit of measure = score) | Pre-surgery to 1, 8, 16, 26, and 52 weeks post-surgery
  Via Patient Reported Outcomes Measurement Information System (PROMIS)
Change in pain (unit of measure = score) | Pre-surgery to 1, 8, 16, 26, and 52 weeks post-surgery
  Via Patient Reported Outcomes Measurement Information System (PROMIS)
Change in depression (unit of measure = score) | Pre-surgery to 1, 8, 16, 26, and 52 weeks post-surgery
  Beck Depression Inventory (BDI II)
Change in fatigue severity (unit of measure = score) | Pre-surgery to 1, 8, 16, 26, and 52 weeks post-surgery
  Fatigue Severity Scale (FSS)

CONTACTS AND LOCATIONS:
Overall Officials: Marcas M Bamman, PhD, Principal Investigator — University of Alabama at Birmingham; S Louis Bridges, MD, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Center for Exercise Medicine, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data might be provided on written request in aggregate form.